CLINICAL TRIAL: NCT01425216
Title: Phase II Trial of Sorafenib in Patients With Extensive Keloids
Brief Title: Sorafenib for Patients With Extensive Keloids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IND application was not approved by the US FDA - Project was never started
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tirgan 11-05
Record Dates: First submitted 2011-08-19; First posted 2011-08-29 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Keloids
Keywords: Keloid; Patient who have extensive or massive keloids
MeSH Terms: conditions — Keloid | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib arm (Experimental): All patients will be treated with sorafenib.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Treatment will be administered on an outpatient basis. All patients will keep a drug diary in order to record compliance with their drug regime. Sorafenib will be taken orally. Maximum length of treatment is 6 months. Starting dose of sorafenib is 200 mg three times per week for one month. In absence of Grade 2 toxicity, the dose will be increased on a monthly basis and will stop at 400 mg twice daily.
  Other Names: Nexavar (sorafenib)

SUMMARY:
Treatment of keloid disorder is an area of unmet medical need. Current treatments for keloid partially address small and localized keloids, yet there are no wholly satisfactory or effective treatments for patients with extensive keloids. Such patients may benefit from effective systemic treatments.

Sorafenib has the potential to regulate the three known dysregulated biological pathways in keloid tissue.

DETAILED DESCRIPTION:
Dysregulation of several intracellular pathways have been reported by various investigators.

[A] Dysregulated apoptosis pathway: p53 mutations have been found in both hypertrophic scar and keloids fibroblasts from cultured cells to various extents. p53 plays a central role in the DNA damage response by inducing cell cycle arrest and/or apoptotic cell death. Time course experiments making cell cultures at different times to investigate the phenomenon of apoptosis and its involvement in the process of pathological scarring in both hypertrophic scars and keloid indicate to dysregulation of apoptotic pathways in Keloid tissue.

[B]Dysregulated TGF- β signaling: Transforming growth factor- β1 (TGF- β1) is well known as the crucial fibrogenic cytokine promoting ECM production and tissue fibrosis in keloid forming [9]. TGF- β1 is an essential profibrotic cytokine for collagen synthesis, and it is well known to increase mRNA expression of procollagen I. Administration of TGF- β1 resulted in a dramatic increase in intracellular collagen I levels in keloid fibroblasts. Due to the close relationship between TGF- β signaling and the production of collagen, blocking TGF- β signaling has the potential of repressing fibroblast proliferation and collagen synthesis, thereby preventing the formation of keloids.

[C]Dysregulated VEGF signaling pathway: VEGF (Vascular endothelial growth factor), one of the most widely studied secreted factors involved in angiogenesis, has been implicated as crucial to normal and pathological wound healing [18]. Gira et al. [19] indicated that VEGF production is abundant in the underlying dermis of keloids. In vitro studies have indicated that VEGF is expressed at higher levels in keloid-derived Fibroblasts than in normal skin Fibroblasts.

Sorafenib is an orally active multikinase inhibitor and has been reported to be an effective inhibitor of apoptosis, TGF-β signaling and VEGF pathway signaling, making it an ideal drug to test in the setting of extensive keloid disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of a keloid.
2. Presence of extensive keloid disease as defined in section 1.3
3. Age 18 to 50
4. A signed informed consent document (ICD)
5. Able and willing to receive sorafenib
6. Patients must have normal end organ and marrow function

Women of child-bearing potential must have a negative pregnancy test during screening. The effects of sorafenib on the developing human fetus are unknown. For this reason, women of child-bearing potential, and men, must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and three months beyond the last dose of sorafenib. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

-

Exclusion Criteria:

1. Diastolic Blood pressure of 90 mm Hg or above
2. History of any degree of hypertension, even medically controlled hypertension
3. History of any form of cardiovascular disease or stroke
4. History of any form of thromboembolic event
5. History of renal dysfunction or proteinuria,
6. History of any form of liver dysfunction
7. History of recent (past 12 month) or planned (next 9 months) major surgery,
8. Men and women who plan to have children within 3 months of their last treatment
9. Psychological Illness that may result in non compliance with treatment
10. Patients receiving any other investigational agents.
11. Patients with a history of serious allergic reactions to eggs (sorafenib is formulated using egg phospholipids).
12. HIV-positive patients receiving combination anti-retroviral therapy are excluded because of possible pharmacokinetic interactions with the investigational agent.
13. Patients who cannot swallow pills for whatever reason will be excluded.
14. Patients having any history or current evidence of a bleeding diathesis.
15. Patients who are taking, or have taken anticoagulants in past 12 months for any reason.
16. Pregnancy and Breast Feeding Pregnant women are excluded from this study because sorafenib has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with sorafenib, breastfeeding is not allowed during the course of the study.

Female patients will be advised not to get pregnant during the first 3 months from last administered dose of sorafenib. Men will be advised to continue using barrier method contraception and not father a child during the first 3 months from last administered dose of sorafenib

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Response Rate (RR) of extensive keloids to sorafenib. RR is the sum of Complete Remission (CR) and Partial Remission (PR) at 12 month after last dose of sorafenib. | 12 months
  The primary objective of this trial is to demonstrate the efficacy of sorafenib in patients with extensive keloids.

SECONDARY OUTCOMES:
The secondary endpoint of this trial is to demonstrate the rate of AE and SAE following exposure to sorafenib measured while on treatment as well as at 1 year after the last dose of sorafenib. | 12 months
  The secondary objective of this trial is to demonstrate safety of sorafenib in this setting. Patients will be followed for one year after their last dose of sorafenib to assess safety of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Principal Investigator — St. Luke's Roosevelt Hospital Center, New York City
Locations (1):
- Michael H. Tirgan, MD, New York, New York, United States